CLINICAL TRIAL: NCT07392697
Title: The Intravenous Amino Acid Therapy for Vascular Rigidity in End Stage Renal Disease
Acronym: NASCAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NASCAR HV
Record Dates: First submitted 2025-09-22; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis; Cardiovascular Calcification
Keywords: carbamylation; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Neither participant nor investigator and outcomes assesor will be aware if patient recived amino acid solution or saline solution. That knowledge will be only available to care provided and coded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amino Acid Supplementation (Experimental): * Product: Synthamin 9® (Baxter), a sterile, pyrogen-free solution of amino acids for injection (5.5%).
  * Dose: 250 ml per administration, providing approximately 13.7 g of free amino acids.
  * Administration: Intravenously during the first hour of hemodialysis.
  * Frequency: Twice weekly (preferably on the two longest HD sessions) for 12 months.
  Interventions: Dietary Supplement: Amino Acid Supplementation
- Placebo (Placebo Comparator): * A sterile, pyrogen-free saline solution
  * Administration: Intravenously during the first hour of hemodialysis.
  * Frequency: Twice weekly (preferably on the two longest HD sessions) for 12 months.
  Interventions: Other: Sterile Saline Arm

INTERVENTIONS:
Dietary Supplement: Amino Acid Supplementation — * Product: Synthamin 9® (Baxter), a sterile, pyrogen-free solution of amino acids for injection (5.5%).
  * Dose: 250 ml per administration, providing approximately 13.7 g of free amino acids.
  * Administration: Intravenously during the first hour of hemodialysis.
  * Frequency: Twice weekly (preferably on the two longest HD sessions) for 12 months.
  Arms: Amino Acid Supplementation
Other: Sterile Saline Arm — Product: Isotonic saline solution (0.9% NaCl), 250 ml.
  • Administration and frequency: Identical to the intervention arm.
  Arms: Placebo

SUMMARY:
The goal of this study is to learn if giving amino acids through the dialysis machine can help protect the blood vessels and heart in people with kidney failure. Patients on dialysis often have problems with stiff blood vessels, which increases their risk of heart attacks, strokes, and other cardiovascular diseases. A chemical change called carbamylation is thought to make blood vessels age and stiffen faster. Amino acids may block this process and improve blood vessel health.

The main questions are:

* Does amino acid treatment reduce the risk of death in dialysis patients?
* Does it improve the health of the heart and blood vessels?
* What side effects or medical problems happen when patients receive amino acids during dialysis?

In this study:

* Participants will be randomly assigned to receive either amino acids (Synthamin 9®) or a placebo (saline).
* The infusion (250 ml) will be given twice a week during dialysis sessions for 12 months.
* After 12 months of treatment, patients will be followed for another 6 months.

During the study, patients will:

* Have regular blood tests to measure markers of blood vessel health, inflammation, and protein carbamylation.
* Undergo heart and vessel tests, including echocardiography, CT scans, and pulse wave velocity measurements.
* Complete quality-of-life questionnaires about symptoms and daily living.

By comparing the amino acid group with the placebo group, researchers will see whether amino acid therapy can make dialysis patients live longer and have healthier hearts and blood vessels.

DETAILED DESCRIPTION:
Background and Rationale Patients with end-stage renal disease (ESRD) who require chronic hemodialysis (HD) face one of the highest cardiovascular mortality rates of any patient population. Despite advances in dialysis technology, medications, and supportive therapies, cardiovascular disease (CVD) accounts for approximately 40-50% of deaths in this group. The excess risk reflects not only traditional risk factors such as hypertension, diabetes, and dyslipidemia but also non-traditional mechanisms that are unique to uremic conditions. Among these, protein carbamylation has emerged as a key biochemical driver of vascular dysfunction and accelerated aging.

Carbamylation is a post-translational modification caused by the reaction of isocyanic acid, a urea-derived metabolite, with free amino groups of proteins. In ESRD, chronically elevated urea concentrations amplify this process. Carbamylation alters structural proteins of the extracellular matrix (collagen, elastin, fibronectin), lipoproteins (LDL, HDL), and clotting factors (fibrinogen, von Willebrand factor), leading to impaired vascular compliance, thrombogenicity, and inflammation. In parallel, carbamylation of endothelial enzymes reduces nitric oxide bioavailability, tipping the balance toward vasoconstriction and hypertension.

Another consequence of carbamylation is the acceleration of cellular senescence. Vascular endothelial and smooth muscle cells exposed to carbamylation undergo growth arrest, increased oxidative stress, and adopt a pro-inflammatory secretory phenotype. Senescent cells amplify vascular inflammation, promote calcification, and further stiffen arteries. Together, these mechanisms establish a vicious cycle of vascular aging in HD patients.

Why Amino Acid Supplementation? During each dialysis session, patients lose 5-12 g of free amino acids into the dialysate. This loss deprives the circulation of natural carbamylation scavengers. Without sufficient free amino acids, reactive isocyanates are more likely to modify proteins. Replacing amino acids intravenously during dialysis directly addresses this imbalance.

* Biochemical rationale: Free amino acids act as competitive substrates for isocyanates, reducing carbamylation of critical structural and functional proteins.
* Physiological rationale: Amino acids, especially arginine, contribute to nitric oxide production, improving vasodilation and endothelial function.
* Clinical evidence: Small pilot studies have shown that amino acid supplementation reduces levels of carbamylated albumin and improves surrogate markers of vascular health. However, no adequately powered randomized trial has tested whether this strategy improves hard outcomes in ESRD.

The NASCAR-PLUS trial (The Intravenous Amino Acid Therapy for Vascular Rigidity in End-Stage Renal Disease) is designed to fill this gap by testing whether intravenous amino acid therapy administered during dialysis can reduce vascular stiffness, improve cardiovascular outcomes, and prolong survival in ESRD patients.

Study Design

The NASCAR-PLUS trial is a multicenter, randomized, double-blind, placebo-controlled clinical trial conducted at five dialysis centers in Norway.

* Population: 104 patients with ESRD undergoing chronic HD or online hemodiafiltration (HDF), on stable treatment regimens for at least 90 days prior to enrollment.
* Randomization: 1:1 allocation to amino acid supplementation or placebo, stratified by site and diabetes status.
* Blinding: Double-blind design, with indistinguishable infusion bags prepared by an unblinded pharmacist.
* Treatment duration: 12 months of intervention, followed by 6 months of observational follow-up.
* Sample size: Powered to detect a clinically meaningful reduction in pulse wave velocity of 0.5 m/s with 80% power at a significance level of 0.05, accounting for dropouts.

Interventions

* Intervention arm: Intravenous Synthamin 9® (Baxter), 250 ml containing 13.7 g amino acids. Administered during the first hour of two weekly dialysis sessions.
* Placebo arm: Intravenous infusion of 0.9% NaCl, 250 ml, under identical conditions.

Infusions are delivered via the venous line of the dialysis circuit. Patients are observed during and after administration for infusion-related reactions.

Clinical Assessments The trial integrates state-of-the-art cardiovascular phenotyping to capture structural, functional, and biochemical effects of the intervention.

Imaging and Functional Assessments

* Pulse Wave Velocity (cf-PWV) and Augmentation Index: Non-invasive gold-standard measures of arterial stiffness performed at baseline, 6 months, and 12 months.
* Coronary Artery Calcium (CAC) Scoring and CT Angiography: Performed at baseline and 12 months to quantify coronary calcification and plaque burden.
* Echocardiography: Comprehensive transthoracic assessments including left ventricular ejection fraction (LVEF), global longitudinal strain (GLS), LV mass, diastolic function (E/e'), and left atrial volume.
* 24-hour Holter ECG: Conducted in a subset of patients at baseline and 12 months to detect arrhythmias and evaluate heart rate variability.

Biomarkers and Biobanking

Blood samples are collected at baseline, months 3, 6, 12, and 18. Analyses include:

* Carbamylation markers: Carbamylated albumin, carbamylated LDL, and free amino acid profiles.
* Inflammation markers: CRP, IL-6, TNF-α, myeloperoxidase.
* Oxidative stress markers: F2-isoprostanes, malondialdehyde, oxidized LDL.
* Vascular injury markers: ICAM-1, VCAM-1, E-selectin.
* Senescence markers: p16^INK4a, p21^CIP1, and senescence-associated secretory phenotype cytokines.

All samples are stored in the Haukeland University Hospital Biobank, creating a long-term research resource for secondary and exploratory studies.

Patient-Reported Outcomes

Quality of life and functional capacity are assessed with validated questionnaires:

* MacNew Heart Disease Health-Related Quality of Life Questionnaire.
* SF-36 Health Survey.
* EQ-5D-5L.

Assessments are performed at baseline, 12 months, and 18 months.

Data Management and Analysis

Data are collected in electronic case report forms (eCRFs) with built-in monitoring and quality checks. All data are anonymized and stored securely in compliance with GDPR and Norwegian data protection laws.

* Primary endpoint analysis: All-cause mortality at 12 months, analyzed with Cox proportional hazards regression, Kaplan-Meier survival curves, and log-rank tests.
* Secondary endpoint analyses: Mixed-effects models for repeated measures (PWV, echocardiography, biomarkers), linear regression for CAC progression, and non-parametric tests for biomarker distributions.
* Subgroup analyses: Pre-specified by diabetes status, baseline inflammation, and dialysis modality.
* Interim analyses: Performed by an independent monitoring board, focusing on safety and feasibility.

Safety Monitoring

Safety is overseen by the clinical investigator team and an independent safety monitoring board. Key elements include:

* Continuous monitoring for infusion-related reactions (hypotension, flushing, nausea, chest discomfort).
* Regular recording of vital signs pre- and post-infusion.
* Adverse events graded according to CTCAE criteria.
* Immediate discontinuation of study drug in cases of serious adverse reaction, with continued safety follow-up.

Patients may withdraw at any time without impact on their standard medical care.

Risk Assessment and Feasibility

The trial builds on strong feasibility data:

* Pilot studies show that amino acid infusions are well tolerated and feasible in the dialysis setting.
* Recruitment is supported by five collaborating centers across Norway, ensuring diversity and robust enrollment.
* Sample size is moderate, but endpoints are designed to capture both survival and mechanistic improvements.

Potential risks include under-recruitment, infusion-related reactions, and dropouts. To mitigate these risks, the trial employs centralized coordination, trained dialysis staff, and standardized operating procedures.

Significance and Impact

If successful, the NASCAR-PLUS trial will provide the first definitive evidence that intravenous amino acid therapy can:

1. Reduce carbamylation and its downstream vascular effects.
2. Improve vascular stiffness and cardiac function in ESRD.
3. Lower mortality and cardiovascular events in a high-risk population.
4. Enhance patient-reported quality of life.

This low-cost, easily implementable therapy could be rapidly integrated into clinical practice worldwide. The mechanistic insights and biobank data will also guide the development of future therapies targeting carbamylation and vascular senescence, with potential relevance not only to kidney disease but also to aging-related cardiovascular and neurodegenerative disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of end-stage renal disease (ESRD) and undergoing maintenance hemodialysis (HD) or online hemodiafiltration (HDF).
* On a stable dialysis regimen for a minimum of 90 consecutive days prior to enrollment.
* Serum albumin level ≥30 g/L.
* Documented dialysis adequacy: single-pool Kt/V (spKt/V) > 1.2.
* Able to understand study procedures and provide written informed consent.

Exclusion Criteria:

* Administration of parenteral amino acids or intravenous nutrition within the past 90 days.
* Severe hypertension (e.g., SBP >180 mmHg despite antihypertensive therapy).
* Advanced liver disease classified as Child-Pugh class C.
* Diagnosis of active malignancy or cancer treatment within the last 5 years.
* Current participation in another interventional study or within the past 30 days.
* Pregnant or breastfeeding women.
* Psychiatric or cognitive impairment that interferes with informed consent or study compliance.
* Life expectancy <12 months due to unrelated comorbidities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality over a 12-month period. | 12 month from enrollment
  This outcome is selected due to the low sample size in each group and the expectation that there may not be many hard cardiovascular events within the 1-year follow-up. The use of all-cause mortality provides a robust endpoint that captures overall patient survival. data will be analyzed with Cox proportional hazard regression, Kaplan -Mayer survival curves and log rank test.

SECONDARY OUTCOMES:
CVD | 12 months from enrollment
  Composite endpoints (MACCE), including heart failure-related hospitalizations, stroke, myocardial infarction, PCI/CABG, and peripheral vascular events. These composite endpoints are designed to assess the broader impact of amino acid therapy on major adverse cardiovascular and cerebrovascular events, providing a comprehensive overview of its effects on cardiovascular outcomes.
CVD 2 - PWV | 12 months from enrollment
  Change in vascular stiffness over a 12-month period, assessed by pulse wave velocity (PWV). The measure of PWV (cartoid to femoral artery) will be measured and compared to reference valus for patients age and sex. These measures will provide a direct assessment of arterial stiffness and vascular compliance, critical indicators of cardiovascular health in ESRD patients
CVD - Alx | 12 months from enrollment
  Change in vascular stiffness over a 12-month period will be assessed by augmentation index (AIx) to provide a direct assessment of arterial stiffness and vascular compliance, critical indicators of cardiovascular health in ESRD patients. The score will be calculated by dividing the augmentation pressure by pulse pressure multiplied by 100.
CVD 3 - CAC | 12 months from enrollment
  Coronary artery calcification (CAC) will be evaluated by the Agatston score, assessed via non-contrast heart CT scans at baseline and the end of the 12-month period. The radiologist will identify areas of calcium in the coronary arteries, multiply the area by a density weighting factor based on Hounsfield density measurements. The score will be presented as 0- low risk; 1-99- Mildly increased risk; 100-299 Moderatly increased risk and 300+ and severly increased risk. This will enable us to evaluate the impact of amino acid therapy on the progression of calcification and atherosclerosis, a major risk factor for CV events in CKD patients
CVD 4 - SIS | 12 months from enrollment
  At baseline and the end of the 12-month period investigators will perform CT coronary angiographies for the identification of coronary stenoses and plaque burden as assessed by the segment involvement score (SIS) on a scale from 1-16
Biomarkers - carbamylation | 12 months from enrollment
  Levels of carbamylated proteins (mg/dl) will be measured at baseline, 6 months, and 12 months. These biomarkers will help elucidate the biological mechanisms through which amino acid therapy may reduce vascular damage and improve cardiovascular outcomes by mitigating carbamylation-induced senescence and promoting endothelial health.
Biomarkers - nitric oxide | 12 months from enrollment]
  Levels of nitric oxide metabolites (nM) will be measured at baseline, 6 months, and 12 months
Biomarkers - cytokines | 12 months from enrollment
  Levels ofinflammatory cytokines (IL-6 - ng/l and TNF-alpha ng/lwill be measured at baseline, 6 months, and 12 months. These biomarkers will help elucidate the biological mechanisms through which amino acid therapy may reduce vascular damage and improve cardiovascular outcomes by mitigating carbamylation-induced senescence and promoting endothelial health.

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland Central Hospital, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
At the moment due to the security reasons (patient data) we dont plan to share idividual patient data. However on request and after vetting in the procedure accepted by the institution the IPD sharing is possible.